CLINICAL TRIAL: NCT07198191
Title: Impact of Sodium-Glucose Cotransporter 2 (SGLT2) Inhibitor Use After Acute Myocardial Infarction in Patients With Type 2 Diabetes: A Nationwide Population Cohort Study
Brief Title: SGLT2 Inhibitor Use After Acute Myocardial Infarction in Patients With Type 2 Diabetes: A Nationwide Cohort Study
Acronym: SGLT2i-AMI
Status: Active, not recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Collaborators: Chong Kun Dang Pharmaceutical Corp. (Industry); Health Insurance Review & Assessment Service (Unknown)
Responsible Party: Principal Investigator, Yongcheol Kim, Principal Investigator, Yonsei University
Other Study IDs: IRB No. 9-2023-0049
Record Dates: First submitted 2025-08-26; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Acute Myocardial Infarction (AMI); Type 2 Diabetes Mellitus (T2DM)
Keywords: SGLT2 inhibitor; Dapagliflozin; Empagliflozin; DPP4 inhibitor; Cardiovascular Outcomes; Heart Failure; Real-world Evidence; NHIS; South Korea
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Heart Failure | interventions — Sodium-Glucose Transporter 2 Inhibitors; dapagliflozin; empagliflozin; Dipeptidyl-Peptidase IV Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SGLT2 Inhibitor Group: Patients with type 2 diabetes mellitus (T2DM) who were prescribed SGLT2 inhibitors after acute myocardial infarction.
  Interventions: Drug: SGLT2 inhibitors (e.g., dapagliflozin, empagliflozin)
- DPP4 Inhibitor Group: Patients with type 2 diabetes mellitus (T2DM) who were prescribed DPP4 inhibitors after acute myocardial infarction.
  Interventions: Drug: DPP4 inhibitors

INTERVENTIONS:
Drug: SGLT2 inhibitors (e.g., dapagliflozin, empagliflozin) — Exposure to SGLT2 inhibitors following AMI in patients with T2DM
  Groups: SGLT2 Inhibitor Group
Drug: DPP4 inhibitors — Exposure to DPP4 inhibitors following AMI in patients with T2DM
  Groups: DPP4 Inhibitor Group

SUMMARY:
This observational, retrospective cohort study aims to evaluate the impact of sodium-glucose cotransporter 2 (SGLT2) inhibitor use after acute myocardial infarction (AMI) in patients with type 2 diabetes mellitus (T2DM). Using the nationwide database from the Korean National Health Insurance Service, the investigators will compare cardiovascular outcomes between patients treated with SGLT2 inhibitors and those treated with dipeptidyl peptidase-4 (DPP4) inhibitors after AMI. The study period includes patients diagnosed with AMI between September 2014 and June 2021, with follow-up data available through June 2022. The primary outcomes include major cardiovascular events (death, myocardial infarction, stroke) and bleeding events. This study will provide real-world evidence on the effectiveness and safety of SGLT2 inhibitors in routine clinical practice following AMI among patients with T2DM in Korea.

DETAILED DESCRIPTION:
Sodium-glucose cotransporter 2 (SGLT2) inhibitors have demonstrated substantial cardiovascular benefits in patients with heart failure and chronic kidney disease, independent of glucose-lowering effects. However, their role in patients with acute myocardial infarction (AMI), particularly in the early post-infarction period, has been less clear. Recently, the DAPA-MI and EMPACT-MI randomized controlled trials have provided important insights. In DAPA-MI, approximately 1 year of dapagliflozin therapy in patients with recent AMI improved cardiometabolic outcomes but did not reduce the composite endpoint of cardiovascular death or hospitalization for heart failure compared with placebo. Similarly, in EMPACT-MI, treatment with empagliflozin among high-risk patients following AMI did not significantly lower the risk of first hospitalization for heart failure or all-cause death compared with placebo. These findings highlight the need for complementary large-scale real-world data to further clarify the clinical utility of SGLT2 inhibitors in this population.

This investigator-initiated observational cohort study utilizes de-identified claims data from the Korean National Health Insurance Service (NHIS) to evaluate clinical outcomes associated with SGLT2 inhibitor use in patients with type 2 diabetes mellitus (T2DM) after AMI. The study population includes adult patients (≥19 years) hospitalized with AMI (ICD-10 codes I21-I23) between September 2014 and June 2021. Patients are stratified based on use of SGLT2 inhibitors versus dipeptidyl peptidase-4 (DPP4) inhibitors following the index event. Exclusion criteria include prior SGLT2 inhibitor use within 12 months before AMI, malignancy, cardiogenic shock, or missing ICD-10 data.

Outcomes of interest include major adverse cardiovascular events (all-cause mortality, cardiovascular death, recurrent MI, ischemic stroke) and bleeding events (major bleeding, site-specific bleeding, transfusion). Propensity-score matching is performed to adjust for baseline demographic and clinical characteristics. Kaplan-Meier survival curves and Cox proportional hazards models are used to estimate hazard ratios for outcomes.

The primary endpoint is the incidence of major adverse cardiovascular events (MACE). Secondary endpoints include individual cardiovascular events, hospitalization for heart failure, and bleeding events. Subgroup analyses assess outcomes according to comorbid chronic heart failure, chronic kidney disease, and concomitant thiazolidinedione therapy.

This study provides real-world evidence on the effectiveness and safety of SGLT2 inhibitors in routine clinical practice following AMI among patients with T2DM in Korea, thereby complementing randomized trial data and informing guideline recommendations for this high-risk population.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥19 years
* Hospitalization with a primary diagnosis of acute myocardial infarction between September 2014 and June 2021
* Diagnosis of type 2 diabetes mellitus (T2DM)
* Prescription of either an SGLT2 inhibitor or a DPP4 inhibitor after index AMI

Exclusion Criteria:

* Diagnosis of type 1 diabetes mellitus
* Gestational diabetes mellitus
* End-stage renal disease (ESRD) or history of kidney transplantation
* No use of either SGLT2 inhibitor or DPP4 inhibitor after index AMI
* Short-term use of SGLT2 inhibitor or DPP4 inhibitor (less than 30 days)
* Concomitant use of SGLT2 inhibitor and DPP4 inhibitor
* Incomplete or missing data for key study variables

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥19 years) with type 2 diabetes mellitus who were hospitalized for acute myocardial infarction in South Korea between September 2014 and June 2021. Eligible patients were identified from the Korean National Health Insurance Service database, with follow-up available through June 2022.
Sampling Method: Non-Probability Sample
Enrollment: 200000 (Estimated)
Dates: Start 2014-09-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Major Adverse Cardiovascular Events (MACE) | From index date (hospitalization for AMI), upto 365 days
  MACE defined as a composite of cardiovascular death, non-fatal myocardial infarction, and non-fatal ischemic stroke.

SECONDARY OUTCOMES:
Incidence of Cardiovascular Death | From index hospitalization for acute myocardial infarction, upto 365 days
  Death from cardiovascular causes, including sudden cardiac death, myocardial infarction, heart failure, or stroke.
Incidence of All-cause Death | From index hospitalization for acute myocardial infarction, upto 365 days
  Death from any cause during follow-up.
Incidence of Non-fatal Myocardial Infarction | From index hospitalization for acute myocardial infarction, upto 365 days
  Hospitalization with a primary diagnosis of myocardial infarction (ICD-10 I21-I22), excluding fatal events.
Incidence of Non-fatal Ischemic Stroke | From index hospitalization for acute myocardial infarction, upto 365 days
  Hospitalization with a primary diagnosis of ischemic stroke, excluding fatal events.
Incidence of Hospital Admission for Heart Failure | From index hospitalization for acute myocardial infarction, upto 365 days
  Hospitalization with a primary diagnosis of heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Yongcheol Kim, MD, PhD, Principal Investigator — Yonsei University Health System, Yongin Severance Hospital
Locations (1):
- Yongin Severance Hospital, Yonsei University Health System, Yongin, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No
The study uses de-identified claims data from the Korean National Health Insurance Service (NHIS). Individual participant data cannot be shared because data access is restricted by NHIS regulations.